CLINICAL TRIAL: NCT06445634
Title: Outcome of Gonioscopy-Assisted Transluminal Trabeculotomy Combined With Goniosynechiolysis in Glaucoma Patients With Secondary Synechial Angle Closure: A Prospective Case Series
Brief Title: Outcome of GATT Combined With Goniosynechiolysis in Glaucoma Patients With Secondary Synechial Angle Closure.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rokaya Emad Radwan, principal investigator, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: _MD-393-2023_
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Glaucoma, Angle-Closure
Keywords: secodary angle closure; GATT; intra ocular pressure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Intervention Model Description: prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gatt combined with goinosynechiolysis in secondary synechial angle closure (Other): Outcome of Gonioscopy-Assisted Transluminal Trabeculotomy Combined with Goniosynechiolysis in Glaucoma Patients with Secondary Synechial Angle Closure
  Interventions: Other: Gonioscopy-Assisted Transluminal Trabeculotomy Combined with Goniosynechiolysis

INTERVENTIONS:
Other: Gonioscopy-Assisted Transluminal Trabeculotomy Combined with Goniosynechiolysis — Gonioscopy-Assisted Transluminal Trabeculotomy Combined with Goniosynechiolysis in Glaucoma Patients with Secondary Synechial Angle Closure
  Other Names: GATT

SUMMARY:
To evaluate the intraocular pressure reduction effect of combined gonioscopy-assisted transluminal trabeculotomy (GATT) with goniosynechialysis in eyes with secondary synechial angle closure glaucoma.

DETAILED DESCRIPTION:
Glaucoma is a group of diseases that present with cupping of the optic nerve head and visual-field defects. It is the most common cause of irreversible blindness all over the world.Angle-closure glaucoma is a type of glaucoma characterized by narrowing or closure of the anterior chamber angle.

Two major types of angle closure glaucoma are defined by the mechanism of angle closure: in appositional contact, the iris is pushed by a pressure difference between the posterior and anterior chambers due to relative pupillary block, while in synechial contact, the peripheral iris adheres to the trabecular meshwork by peripheral anterior synechiae (PAS). PAS can develop in various ocular conditions, including: ocular inflammation, a post-traumatic condition, after cataract surgery, or with an iris bombe in a pupillary block glaucoma.

Grover et al. described a technique for ab-Interno circumferential trabeculotomy termed gonioscopy-assisted transluminal trabeculotomy (GATT). The procedure aims to create a 360° trabeculotomy from an ab-Interno approach.

GATT procedure is a MIGS technique in which trabecular meshwork is circumferentially bypassed by incising it using a suture or microcatheter.In this technique, aqueous humor passes through the collector channels and episcleral veins through the cleaved open diseased trabecular meshwork.

Elsayed et al previously demonstrated that combining phacoemulsification with GATT in PACG yielded more favorable outcomes in terms of IOP, glaucoma medications and surgical success compared to phacoemulsification alone.However, to date, no studies have looked at the outcomes of combining goniosynechialysis with GATT in secondary angle closure glaucoma. In fact, most studies looking at the outcomes of GATT in different types of glaucoma excluded eyes with synechial angle closure.

Goniosynechialysis (GSL) is the process of physically separating PAS, which can develop in the trabecular meshwork due to various conditions including primary and secondary cases of angle closure.

So, for those cases of synechial angle closure glaucoma combining GATT and GSL might aid in the IOP lowering effect required.

ELIGIBILITY:
Inclusion Criteria:

* Patients with secondary synechial angle closure glaucoma
* Involving more than 180 degrees of the iridocorneal angle
* Requiring surgery for uncontrolled IOP despite maximum tolerated therapy.

Exclusion Criteria:

* Eyes with PACG.
* Eyes with neovascular glaucoma. (Some apparently stable NVG cases would have remnants of neo-vessels in the angle that are hidden behind the synechiae).
* Eyes with retinal pathology.
* Eyes requiring combined phacoemulsification and GATT.
* Eyes with corneal pathology that can preclude surgery and imaging.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
IOP and glaucoma medications. | 1day,1 week,1 months, 3 months, 6 months and 1 year
  measurement of intra ocular pressure and documentation of number of anti glaucoma medications post operative
Surgical success. | 1day,1 week,1 months, 3 months, 6 months and 1 year
  Surgical success will be defined as: complete if IOP is less than or equal to 21mmHg without medications and qualified success if IOP is less than or equal to 21mmHg with medications. Failure will be the inability to achieve such a pressure, the need for another glaucoma operation or the development of a sight-threatening complication (e.g., retinal detachment, endophthalmitis)

SECONDARY OUTCOMES:
Complications. | 1day,1 week,1 months, 3 months, 6 months and 1 year
  rate of complications will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy Hospitals, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
medical data including intraocular pressure and study outcomes will be shared but excluding any participant confidential data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication within 18 months
Access Criteria: will be uploaded